CLINICAL TRIAL: NCT05239884
Title: CSD201202: A Randomized, Crossover, Confinement Study to Assess Nicotine Uptake From Electronic Nicotine Delivery System P12
Brief Title: CSD201202: A Study to Assess Nicotine Uptake From Electronic Nicotine Delivery System P12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD201202
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Smoking; Tobacco Use
MeSH Terms: conditions — Smoking; Tobacco Use | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Product usage order EFDGCHBA (Experimental): Subjects will use each of the 8 products (EFDGCHBA) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: ENDS Product A with 1.5% nicotine; Other: ENDS Product B with 1.5% nicotine; Other: ENDS Product C with 1.5% nicotine; Other: ENDS Product D with 1.5% nicotine; Other: ENDS Product E with 1.5% nicotine; Other: ENDS Product F with 1.5% nicotine; Other: ENDS Product G with 1.5% nicotine; Other: ENDS Product H with 1.5% nicotine
- Product usage order HAGBFCED (Experimental): Subjects will use each of the 8 products (HAGBFCED) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: ENDS Product A with 1.5% nicotine; Other: ENDS Product B with 1.5% nicotine; Other: ENDS Product C with 1.5% nicotine; Other: ENDS Product D with 1.5% nicotine; Other: ENDS Product E with 1.5% nicotine; Other: ENDS Product F with 1.5% nicotine; Other: ENDS Product G with 1.5% nicotine; Other: ENDS Product H with 1.5% nicotine
- Product usage order CDBEAFHG (Experimental): Subjects will use each of the 8 products (CDBEAFHG) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: ENDS Product A with 1.5% nicotine; Other: ENDS Product B with 1.5% nicotine; Other: ENDS Product C with 1.5% nicotine; Other: ENDS Product D with 1.5% nicotine; Other: ENDS Product E with 1.5% nicotine; Other: ENDS Product F with 1.5% nicotine; Other: ENDS Product G with 1.5% nicotine; Other: ENDS Product H with 1.5% nicotine
- Product usage order DECFBGAH (Experimental): Subjects will use each of the 8 products (DECFBGAH) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: ENDS Product A with 1.5% nicotine; Other: ENDS Product B with 1.5% nicotine; Other: ENDS Product C with 1.5% nicotine; Other: ENDS Product D with 1.5% nicotine; Other: ENDS Product E with 1.5% nicotine; Other: ENDS Product F with 1.5% nicotine; Other: ENDS Product G with 1.5% nicotine; Other: ENDS Product H with 1.5% nicotine
- Product usage order FGEHDACB (Experimental): Subjects will use each of the 8 products (FGEHDACB) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: ENDS Product A with 1.5% nicotine; Other: ENDS Product B with 1.5% nicotine; Other: ENDS Product C with 1.5% nicotine; Other: ENDS Product D with 1.5% nicotine; Other: ENDS Product E with 1.5% nicotine; Other: ENDS Product F with 1.5% nicotine; Other: ENDS Product G with 1.5% nicotine; Other: ENDS Product H with 1.5% nicotine
- Product usage order BCADHEGF (Experimental): Subjects will use each of the 8 products (BCADHEGF) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: ENDS Product A with 1.5% nicotine; Other: ENDS Product B with 1.5% nicotine; Other: ENDS Product C with 1.5% nicotine; Other: ENDS Product D with 1.5% nicotine; Other: ENDS Product E with 1.5% nicotine; Other: ENDS Product F with 1.5% nicotine; Other: ENDS Product G with 1.5% nicotine; Other: ENDS Product H with 1.5% nicotine
- Product usage order ABHCGDFE (Experimental): Subjects will use each of the 8 products (ABHCGDFE) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: ENDS Product A with 1.5% nicotine; Other: ENDS Product B with 1.5% nicotine; Other: ENDS Product C with 1.5% nicotine; Other: ENDS Product D with 1.5% nicotine; Other: ENDS Product E with 1.5% nicotine; Other: ENDS Product F with 1.5% nicotine; Other: ENDS Product G with 1.5% nicotine; Other: ENDS Product H with 1.5% nicotine
- Product usage order GHFAEBDC (Experimental): Subjects will use each of the 8 products (GHFAEBDC) during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: ENDS Product A with 1.5% nicotine; Other: ENDS Product B with 1.5% nicotine; Other: ENDS Product C with 1.5% nicotine; Other: ENDS Product D with 1.5% nicotine; Other: ENDS Product E with 1.5% nicotine; Other: ENDS Product F with 1.5% nicotine; Other: ENDS Product G with 1.5% nicotine; Other: ENDS Product H with 1.5% nicotine

INTERVENTIONS:
Other: ENDS Product A with 1.5% nicotine — P1211216, an Electronic Nicotine Delivery System (ENDS) with 1.5% nicotine
Other: ENDS Product B with 1.5% nicotine — P1213516, an Electronic Nicotine Delivery System (ENDS) with 1.5% nicotine
Other: ENDS Product C with 1.5% nicotine — P1213416, an Electronic Nicotine Delivery System (ENDS) with 1.5% nicotine
Other: ENDS Product D with 1.5% nicotine — P1212716, an Electronic Nicotine Delivery System (ENDS) with 1.5% nicotine
Other: ENDS Product E with 1.5% nicotine — P1213716, an Electronic Nicotine Delivery System (ENDS) with 1.5% nicotine
Other: ENDS Product F with 1.5% nicotine — P1213816, an Electronic Nicotine Delivery System (ENDS) with 1.5% nicotine
Other: ENDS Product G with 1.5% nicotine — P1211916, an Electronic Nicotine Delivery System (ENDS) with 1.5% nicotine
Other: ENDS Product H with 1.5% nicotine — P1210016, an Electronic Nicotine Delivery System (ENDS) with 1.5% nicotine

SUMMARY:
This is an open-label, randomized, 8-way crossover study designed to evaluate plasma nicotine pharmacokinetic (PK) parameters following an ad libitum use of Electronic Nicotine Delivery System (ENDS) investigational products (IPs) in a confinement setting by generally healthy combustible cigarette (CC) smokers and dual users of CC and ENDS.

DETAILED DESCRIPTION:
This study is designed to evaluate plasma nicotine pharmacokinetic (PK) parameters following the use of Electronic Nicotine Delivery System (ENDS) investigational products (IPs) in generally healthy combustible cigarette (CC) smokers and dual users of CC and ENDS.

Potential subjects will complete a pre-screening interview and a Screening Visit to assess eligibility within 45 days prior to enrollment, randomization and confinement.

Following the Screening Visit, eligible subjects will be scheduled for a check-in and randomization visit. At the check-in and randomization visit, subjects' continued eligibility will be confirmed prior to being randomized to a product use sequence and beginning 9 nights and 10 days of confinement.

Starting on study Day 1, subjects will start a Pre-study ENDS IP Acclimation Period. During Pre-Study Product Acclimation Period, subjects will be required to acclimate to each of the ENDS IP at least once, while having access to their usual brand (UB) cigarettes for ad libitum use. Starting on Day 3, subjects will participate in eight separate Test Sessions for nicotine PK assessment, one for each ENDS IP. For approximately a half day prior to each respective Test Session (starting on Day 2), subjects will use the assigned ENDS IP for the following day's Test Session at least four times.

Starting on Day 3 and continuing through Day 10, subjects will participate in eight separate Test Sessions, one for each IP that will last for approximately 4 hours following the start of 5 minutes of ad libitum IP use. During each Test Session, subjects will use one of the eight IPs. The ENDS IP for each Test Session will be determined based on a randomly assigned ENDS IP presentation schedule, where an 8-sequence ENDS IP use schedule will be generated using a Williams Design. Each Test Session will be preceded by a 12-hour tobacco/nicotine product abstention the night before.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy male or female, 21 to 60 years of age, inclusive, at the time of consent.
3. Expired breath carbon monoxide level is ≥ 10 ppm and ≤ 100 ppm at Screening.
4. Positive urine cotinine test at Screening.
5. Smokes only combustible filtered, menthol or non-menthol combustible cigarettes (CC), 83 mm to 100 mm in length.
6. Agrees to smoke same usual brand (UB) cigarette throughout the study period. UB cigarette is defined as the cigarette brand style currently smoked most frequently by the subject.
7. Subjects must meet one (a or b) of the following tobacco use conditions:

   1. Smokes at least 10 cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the Principal Investigator (PI).
   2. Dual user of CC and electronic cigarettes (ECs) who self-reports:

   i. Smoking at least 10 cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening Visit. Brief periods of abstinence more than 30 days prior to screening due to illness, quit attempt or clinical study participation will be allowed at the discretion of the Investigator and ii. Using a nicotine-containing electronic nicotine delivery system (ENDS) (cartridge or a tank system).
8. Willing to use only UB cigarette and ENDS during the study period.
9. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to each Test Session.
10. Females must be willing to use a form of contraception acceptable to the PI from the time of signing informed consent until End-of-Study.
11. Agrees to in-clinic confinement of 10 days and 9 nights.

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study subject unsuitable to participate in this clinical study.
2. History, presence of, or clinical laboratory test results indicating diabetes.
3. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95mmHg, measured after being seated for five minutes at Screening and at check-in Day 1.
4. Weight of ≤ 110 pounds.
5. Hemoglobin level is < 12.5 for females or <13.0 for males g/dL at Screening.
6. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion pending approval from the Medical Monitor.
7. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
8. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
9. Must not be a current regular user (i.e., > 5 times per month) of any tobacco products other than CCs or ENDS within the last 6 months prior to screening.
10. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (NRT) (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing of informed consent.
11. History or presence of bleeding or clotting disorders.
12. Any use of anticoagulants or daily use of aspirin (≥ 325 mg).
13. Whole blood donation within 8 weeks (≤ 56 days) prior to the signing of informed consent and between Screening and check-in Day 1.
14. Plasma donation within (≤) 7 days prior to the signing of informed consent and between Screening and check-in Day 1.
15. Participation in another clinical trial within (≤) 30 days prior to the signing of informed consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.
16. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
17. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
18. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening or Day 1.
19. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or a previous quit attempt within (≤) 30 days prior to the signing of the ICF.
20. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol result at Screening or Day 1.
21. Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
22. Determined by the PI to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
AUC nic 0-240 | 0 to 240 minutes
  Baseline-adjusted area under the plasma nicotine concentration-versus-time curve from time zero to 240 minutes after the start of IP use. A relative estimate of nicotine absorption that results from a single use of each of the ENDS IP.
Cmax | 240 minutes
  The maximum plasma concentration of nicotine attained over 240 minutes after the start of ENDS IP use.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hong, MD, Study Director — RAIS
Locations (1):
- High Point Clinical Trials Center, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No